CLINICAL TRIAL: NCT02444182
Title: Effect of Lactobacillus Rhamnosus LGG and Bifidobacterium Lactis BB-12 on Gingival Health and Dental Plaque in Healthy Adolescents: a Randomized Controlled Clinical Trial
Brief Title: Effects of Probiotics on Oral Health
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kuwait University (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, ABRAR ALANZI, ASSISTANT PROFESSOR, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DD04/13
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Periodontal Health; Dental Plaque Accumulation
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): participants will receive a lozenge containing mixture of probiotic bacteria BB-12 and LGG
  Interventions: Dietary Supplement: Probiotics
- Control - No probiotics (Placebo Comparator): Participants will receive a control lozenge containing no probiotics. all lozenges are sugar-free; sweetened by xylitol (0.5 g xylitol per piece)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — A half of the participants will be randomly allocated to the probiotics group. They will receive a probiotics lozenge twice a day for 4 weeks. Pre and Post intervention clinical exam will be conducted
  Arms: Probiotics
Dietary Supplement: Placebo — A half of the participants will be randomly allocated to the placebo group. Lozenges with no probiotics will be given twice daily for 4 weeks. Pre and Post intervention clinical exam will be conducted
  Arms: Control - No probiotics

SUMMARY:
Some probiotics have been shown to have preventive effects on infectious diseases and allergies. Because their long-term enhancement of the immune responses of children, they have been recommended for infants in some countries. The most promising ones seem to be the combination of Bifidobacterium lactis BB-12 and Lactobacillus rhamnosus GG. Probiotic microbes are mainly ingested orally and the gastrointestinal tract is thus the primary target organ for them. However, the mouth is the first part of the gastrointestinal tract. Most probiotics are in theory cariogenic, thus their effects on oral health should be known. Several probiotics decrease levels of salivary mutans streptococci (MS), but in other respects very little is known about their effects on the oral microbiota. Also effects of probiotics on dental plaque should be studied. This study aims to find out the effects of the combination of BB-12 and LGG, delivered with a lozenge (4 weeks, twice a day) with a mixture of them on the amount of plaque and gingival health

DETAILED DESCRIPTION:
The Food and Agriculture Organization (FAO) of the United Nations and the World Health Organization (WHO) have defined probiotics as "live micro-organisms, which when administered in adequate amounts, confer a health benefit to the host" (WHO 2002). They should preferably be of human origin, be able to temporarily colonize the gastrointestinal tract and survive in it. They must also be non-pathogenic and non-toxic.

Probiotics are used in the prevention and treatment of infectious diseases and allergies (Hatakka and Saxelin, 2008; Salminen et al., 2010). In some countries probiotics are recommended for infants and adults because of their long-term enhancement of the immune responses. Combinations of probiotics, like Bifidobacterium lactis BB-12 (BB-12) and Lactobacillus rhamnosus GG (LGG), appear to be most effective in this respect (Isolauri et al., 2000; Rautava et al., 2009; Smith et al., 2012). Probiotics are mainly ingested orally, and the gastrointestinal tract is thus the primary target organ for probiotic micro-organisms. However, when ingested in the form of for example tablets, chewing gums, cheese and milk, the oral cavity is exposed to the probiotics. With the world-wide increase in the use of probiotics their effects of on oral health have become a hot topic.

Many types of probiotic bacteria have been explored but the most widely studied species are those that belong to the genera Lactobacillus and Bifidobacterium. Yogurt and fermented milk products are considered the simplest source of probiotic administration for humans. The proven effects of probiotics in general health has led to more research in the oral health field including dental caries, periodontal disease and halitosis. Some clinical studies have demonstrated a decrease in the cariogenic mutans streptococci counts and in dental plaque (Näse et al. 2001, Ahola et al. 2002, Nikawa et al. 2004, Caglar et al. 2007, Twetman & Keller 2012). Probiotics have also shown improvements in the periodontal status in patients with periodontal disease (Riccia et al. 2007, Shimauchi et al. 2008, Teughels et al. 2013, Yanine et al. 2013). Recently, Toiviainen et al. (2015) found that the combination of Lactobacillus rhamnosus GG (LGG) and Bifidobacterium strain Bifidobacterium lactis (BB-12) improved the periodontal health in healthy adults by reducing the plaque amount and subsequently the gingival inflammation without affecting the oral microbiota.

More evidence is necessary to confirm the efficacy of the combination of LGG and BB-12 in the oral health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adolescent - ASA I & II
* No Antibiotics use
* No intake of commercially available probiotics products during the intervention

Exclusion Criteria:

* Adolescents have ASA III or IV
* Antibiotics use
* refuse to stop taking commercially available probiotics products during intervention

Ages: 13 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABRAR N ALANZI, MS, Principal Investigator — KUWAIT UNIVERISTY
Locations (1):
- Abdullah Alwaheeb intermediate School, Kuwait City, Kuwait, Kuwait

REFERENCES:
- [Result] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Inclusion criteria of the study:
  * healthy subject with no history of systemic antibiotics or topical fluoride treatments within the 4 weeks prior to baseline
  * subject who agrees to suck lozenges containing probiotics twice a day.
  * subject who agrees to stop taking any other probiotic containing products during the study period
Groups:
- Probiotics: participants received a lozenge containing mixture of probiotic bacteria BB-12 and LGG
  Probiotics: A half of the participants was randomly allocated to the probiotics group. They received probiotics lozenges twice a day for 4 weeks. Pre and Post intervention clinical exams were conducted
- Control - No Probiotics: Participants received a control lozenge containing no probiotics. all lozenges were sugar-free; sweetened by xylitol (0.5 g xylitol per piece)
  Placebo: A half of the participants was randomly allocated to the placebo group. Lozenges with no probiotics were given twice daily for 4 weeks. Pre and Post intervention clinical exams were conducted
Period: Overall Study
Arm/Group | Probiotics | Control - No Probiotics
Started | 54 | 54
Completed | 52 | 49
Not Completed | 2 | 5
Not completed — non-compliance | 2 | 1
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: Sample size determination was based on the data by Toiviainen et al. (2015). A sample size of 104 subjects (92 + 10% to provide cover in case of subject drop out) was predicted to provide 80% power with an α of 0.05.
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics | Control - No Probiotics | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] — school children in 7-9th grades (aged 13-15 years)
  years | 14 (1) | 14 (1) | 14 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 54 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 54 | 108
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kuwait | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Gingival Health
Description: The gingival Index of Loe and Silness (1963) was used to record all surfaces (buccal, lingual, mesial, distal) for index teeth (16, 12, 24, 36, 32, 44). Gingival pockets were gently touched with a periodontal probe and possible bleeding was registered.
  The criteria are:
  0 = no inflammation
  1. = mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding
  The GI of the tooth was determined by adding the scores of the four surfaces and divided the total by four.
  The GI of the individual was obtained by adding the values of each tooth and dividing by the number of teeth examined
  A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation, and 2.1-3.0 = severe inflammation
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotics | Control - No Probiotics
Number analyzed (Participants) | 52 | 49
units on a scale | 0.46 (0.6) | 0.18 (0.39)
Statistical Analysis 1: Comparison: Probiotics vs Control - No Probiotics; Null hypothesis was no difference in Gingival index between probiotics and control groups; Test type: Superiority or Other; p = 0.015, paired t-test; Mean Difference (Net) = 0.28, Standard Deviation 0.21

2. Primary Outcome: Plaque Index
Description: A modified Quickley-Hein plaque index (PI) was used to record the buccal and lingual surfaces of all teeth (from right second molar to left second molar) 0 = no plaque
  1. = separate flecks of plaque at the cervical margin of the tooth
  2. = a thin continuous band of plaque at the cervical margin
  3. = a band of plaque wider than 1 mm but covering less than 1/3 of the crown
  4. = plaque covering at least 1/3 but less than 2/3 of the crown
  5. = plaque covering 2/3 or more of crown
  An index for the entire mouth is determined by dividing the total score by the number surfaces (a maximum of 2 x 2 x 14 = 56 surfaces) examined.
  ** Plaque index score reported in the table below represents Pl for the entire mouth. the range is between 0 (no plaque) to 5 (maximum plaque coverage)
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Probiotics | Control - No Probiotics
Number analyzed (Participants) | 52 | 49
units on a scale | 0.80 (0.76) | 0.71 (0.67)
Statistical Analysis 1: Comparison: Probiotics vs Control - No Probiotics; Null hypothesis was no difference in plaque index between probiotics and control groups; Test type: Superiority or Other; p = 0.909, paired t-test; Mean Difference (Final Values) = 0.09, Standard Deviation 0.09

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Probiotics | Control - No Probiotics
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

LIMITATIONS AND CAVEATS:
limitations of this study include:

1. short period: only 4 weeks to reach maximum compliance
2. number of participants: just above the minimum sample size due to refusal of many parents to give consent for their children participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No